CLINICAL TRIAL: NCT06573112
Title: Incidence, Factors Associated and Outcomes of Central Venous Catheter-Related Thrombosis in Critically Ill Patients, a Prospective Cohort Study
Brief Title: Central Venous Catheter-Related Thrombosis in Critically Ill Patients
Acronym: CVC-RT
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr Jyoti Burad, Senior Specialist, Sultan Qaboos University
Other Study IDs: #3299
Record Dates: First submitted 2024-08-01; First posted 2024-08-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-08

CONDITIONS: Catheter Related Complication
Keywords: central venous catheter thrombosis; incidence; complications; length of stay
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cetral venous catheter group: ICU patients with a new central venous catheter.
  Interventions: Diagnostic Test: ultrasound assessment for catheter-related thrombosis.

INTERVENTIONS:
Diagnostic Test: ultrasound assessment for catheter-related thrombosis. — Patients with newly inserted central venous catheter will be assessed with vascular ultrasound for the presence of catheter-related thrombosis

SUMMARY:
This project aims to identify catheter-related thrombosis (CRT) and determine its incidence, associated factors, and outcomes. The eligible patients will undergo daily ultrasound just distal to the central venous catheter insertion site for CRT. A staff radiologist will review all positive cases. These cases will be monitored by daily ultrasound examination till three days after the removal of the catheter or till the patient stays in the intensive care unit (ICU). The patient demographics, ICU treatment details, and outcomes will be noted. The data will be then analyzed. A preventive strategy will be prepared and disseminated to the department personnel to improve the quality of care.

DETAILED DESCRIPTION:
Central venous catheter (CVC) insertion is a common procedure for critically ill patients. The CVCs are inserted on any site, including the internal jugular, subclavian, brachio-cephalic, and femoral veins. The endothelium of the vein is injured with CVC placements, and this predisposes to the formation of thrombus in addition to other predisposing factors like immobility, thrombophilia, reduced venous blood flow, hypercoagulable state, catheter material, catheter diameter to vein diameter ratio, CVC tip position, etc. The catheter fills up the lumen space intravenously, thereby reducing blood flow inside the vein. This slow flow state can predispose to thrombus formation.

Peripherally inserted central catheters might have a higher incidence of CRT due to this reason. CRT forms mostly at the insertion site, frequently within the first week of catheterization. The clinical manifestation of CRT can vary according to the size and site of the thrombus. It is frequently asymptomatic; however, most patients develop signs and symptoms like edema, pain, erythema, weakness, and sometimes superficial venous circles (Urschel's sign). If the vein involved with CRT is the superior vena cava of the anonymous vein, there could be signs of superior vena cava (SVC) syndrome. CRT is frequently evident with inadequate catheter flow. As a consequence of CVC thrombus development at different sites and severity, complications like deep vein thrombosis (DVT) extension, compartment syndrome, SVC syndrome, catheter infection, and permanent venous obstruction can develop. Sometimes, there can be the end-organ effect of the thrombus migration, causing a pulmonary embolism (PE), ischemic stroke, and embolism to the gut, liver, kidneys, and heart. These can significantly impact the patient outcome, such as the length of stay in the ICU.

Aim of the Study: This research aims to study the incidence and associated factors, including the initial catheter-to-vein diameter ratio, and the outcomes of CRT at a tertiary-level university hospital in Oman. With these data, we will understand the condition and form a preventive strategy for CRT for critically ill patients.

Methods: This prospective study will include enrollment, daily observation, and follow-up of all patients undergoing a new CVC placement in the ICU. After obtaining ethical approval, the study will be registered at one of the registries (Clinicaltrials platform). All patients admitted to the ICU would be approached, and those getting CVC placement would be given information about this research with the help of an information sheet. All patients/or their relatives who consent to participate will be included during the study period. Ultrasound assessment will be done on admission and every day till discharge from ICU or up to three days after CVC removal if in ICU.

Ultrasound assessment: This will involve examination of the central vein at and distal to the catheter site. The examination will detect echogenic mass and compressibility in the vein, as well as evaluate the color flow. A diagnosis of CRT will be made if there is an echogenic mass and either incompressibility or absent color flow. A radiologist will review all the positive cases. Partial occlusion will be defined by partially occluding intraluminal echogenic filling defect, and complete occlusion will be defined as intraluminal occluding thrombus with rounding and non-compressibility of vein and absence of color flow on Doppler. In addition to the diagnosis, the dimensions of the thrombus will be measured every day. The outer diameter of the catheter and the catheter-vein diameter (CVD) ratio will be calculated on the day of CVC insertion. The extraluminal hematoma will also be measured.

Data collection: Data like patient demographics, co-morbidities, severity of illness SOFA (sequential organ failure assessment) score, investigations (hemoglobin level, platelet counts, coagulation profile, liver and renal dysfunction, plasma protein levels, calcium levels, blood group etc.), catheterization details (site and side of catheterization, number of venous puncture attempt, peri-venous hematoma/collection, CVD ratio at the start, compressibility, rounding of vein, presence of color doppler flow), treatment (medications like antibiotics, antiplatelets, pro- thrombotic medications like tranexamic acid, factor 7a, vitamin D, vitamin K, intravenous immunoglobulin; other regular ICU prophylaxis like DVT prophylaxis with unfractionated and fractionated heparin or other medications, peptic ulcer prophylaxis with proton pump blockers, medication/total parenteral nutrition with high osmolality etc.) in ICU. Other routine ICU treatments with extracorporeal machines like continuous renal replacement therapy(CRRT), extracorporeal membrane oxygenation (ECMO), plasmapheresis, intermittent hemodialysis; length of stay in ICU, outcomes like end organ thrombosis like ischemic stroke, renal/hepatic/splenic/gut/myocardial infarction etc. will be recorded prospectively in ICU and from electronic patient records from hospital information system after the discharge from ICU till hospital stay of the patient. The ICU course record will also include the treatment procedures, ventilator days, infection details, especially the catheter-related bloodstream infections, and radiological assessment of the position of the tip of the catheter will all be recorded.

Sample size:

The sample size was estimated based on the anticipated cumulative incidence of CRT in an ICU population (primary outcome). The literature showed that the incidence ranges from 15-20%. We expect around 500 ICU patients to be catheterized during the study period. We anticipated a CRT incidence of 17% with a 3% absolute precision. The confidence level was set at 95%. Therefore, the researcher has to study at least 274 admitted catheterized patients in the ICU. The sample size was calculated using the OpenEpi web application (https://www.openepi.com/SampleSize/SSPropor.htm).

Statistical analysis Continuous variables will be presented as mean, median, standard deviation, and interquartile range, whereas categorical variables will be presented as frequency and percentage. The comparison of means between the two groups will be assessed using the independent samples t-test between two categorical variables will be tested using a Chi-square test (Fisher's exact/Likelihood ratio). The cumulative incidence of CRT will be reported with its 95% CI. CRT incidence rate and 95% CI will be expressed as events/1000 catheter days. Univariate and multivariate Cox proportional hazards regression models will be fitted to calculate hazard ratios (HR) and 95% CI of CRT. A P-value less than 0.05 will be considered statistically significant. All the analyses will be performed using IBM SPSS Statistics (IBM Corp. Released 2022. IBM SPSS Statistics for Windows, Version 29.0. Armonk, NY: IBM Corp).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) undergoing Central Venous Catheter (CVC) placements in the ICU or emergency department while waiting for admission to the ICU.

Exclusion Criteria:

* Pre-existing deep vein thrombosis (DVT),
* Pre-existing CVC at ICU admission (other than placement in the emergency department)
* Refusal to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (>18 years) admitted to the ICU who receive a new CVC placement in the ICU or just before admission to the ICU in the emergency department of the tertiary hospital specified will be considered potential candidates for the study. Once they fulfill the inclusion criteria, those whose surrogates or patients themselves consent to the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2024-07-21 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Catheter-related thrombosis (CRT) | one year approximately
  Incidence of CRT in critically ill patients

SECONDARY OUTCOMES:
Rate of cases developing ischemic complications | one year approximately
  Rate of new onset of myocardial infarction (diagnosis by electrocardiogram [ECG] + troponin), stroke, gut ischemia, spleen, liver, and kidney infarction (diagnosis by computerized tomography [CT] scan)
Presence of factors associated with the development of CRT | one year approximately
  Association of presence of various factors with the development of CRT (measured by uni- and multivariate regression analysis) like demographics (age>60 years, gender), co-morbidities (diabetes, hypertension, heart disease, chronic obstructive pulmonary disease, stroke, kidney failure, lymphoma/leukemia, sickle cell disease), treatment modalities (medications: antibiotics, thrombogenic medications, hyper-osmolar medications; derangement in lab values like thrombocytosis, polycythemia, plasma albumin level [g/dl] above or below normal range, presence/absence of deep vein thrombosis prophylaxis; ventilation days more than 7 days) extracorporeal therapies (presence/absence of dialysis, plasmapheresis, and extracorporeal membrane oxygenation), and catheter-related factors like catheter-vein diameter ratio more than 33% and number of catheter days more than 10 days
Mortality at 28 and 90 days | one year approximately
  Mortality at 28 and 90 days till hospital discharge
Length of stay in ICU | one year approximately
  Length of stay in ICU for each episode of ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, MD EDIC FICM, Principal Investigator — Sultan Qaboos University Hospital, University Medical City
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Muḩāfaz̧at Masqaţ, Oman

IPD SHARING:
Plan to Share IPD: Undecided
IPD might be shared without patient identity after publication if the interested party contacts the principle investigator

REFERENCES:
- [Background] Geerts W. Central venous catheter-related thrombosis. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):306-11. doi: 10.1182/asheducation-2014.1.306. Epub 2014 Nov 18. PMID 25696870
- [Background] Evans NS, Ratchford EV. Catheter-related venous thrombosis. Vasc Med. 2018 Aug;23(4):411-413. doi: 10.1177/1358863X18779695. Epub 2018 Jun 28. No abstract available. PMID 29952254
- [Background] Wu C, Zhang M, Gu W, Wang C, Zheng X, Zhang J, Zhang X, Lv S, He X, Shen X, Wei W, Wang G, Lu Y, Chen Q, Shan R, Wang L, Wu F, Shen T, Shao X, Cai J, Tao F, Cai H, Lu Q; Study Group of Central Venous Catheter-related Thrombosis. Daily point-of-care ultrasound-assessment of central venous catheter-related thrombosis in critically ill patients: a prospective multicenter study. Intensive Care Med. 2023 Apr;49(4):401-410. doi: 10.1007/s00134-023-07006-x. Epub 2023 Mar 9. PMID 36892598
- [Background] Andrews K, Fitzgerald M. Cutaneous flexion reflex in human neonates: a quantitative study of threshold and stimulus-response characteristics after single and repeated stimuli. Dev Med Child Neurol. 1999 Oct;41(10):696-703. doi: 10.1017/s0012162299001425. PMID 10587047
- [Background] Grant JD, Stevens SM, Woller SC, Lee EW, Kee ST, Liu DM, Lohan DG, Elliott CG. Diagnosis and management of upper extremity deep-vein thrombosis in adults. Thromb Haemost. 2012 Dec;108(6):1097-108. doi: 10.1160/TH12-05-0352. Epub 2012 Oct 23. PMID 23093319
- [Background] Linenberger ML. Catheter-related thrombosis: risks, diagnosis, and management. J Natl Compr Canc Netw. 2006 Oct;4(9):889-901. doi: 10.6004/jnccn.2006.0074. PMID 17020667
- [Background] Raziuddin S, Elawad ME, Benjamin B. T-cell abnormalities in antibody deficiency syndromes. Scand J Immunol. 1989 Oct;30(4):419-24. doi: 10.1111/j.1365-3083.1989.tb02445.x. PMID 2814365